CLINICAL TRIAL: NCT04785703
Title: Prolactin Hormone in Oral Lichen Planus Tissue Samples
Brief Title: Prolactin Hormone in Oral Lichen Planus
Status: Completed | Type: Observational
Sponsor: October University for Modern Sciences and Arts (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Naglaa Elwakeel, professor, October University for Modern Sciences and Arts
Other Study IDs: REC18-048
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- oral lichen planus group: patients with chronic bollus erosive lichen planus

SUMMARY:
Oral lichen planus (OLP) is one of the most common mucosal diseases with autoimmune etio-pathogenesis with involvement of various cytokines similar to psoriasis.It generally occurs more commonly in females, in a ratio of 3:2. prolactin (PRL),It is a peptide hormone that has a role in autoimmune related diseases like systemic lupus erythematosus and , rheumatoid Artheritis. The role of PrL in OLP pathogenesis was never investigated.the aim of this study is to investigate the expression of PRL receptors in tissue biopsies of OLP patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with oral lichen planus
* systemically healthy

Exclusion Criteria:

* oral lichenoid lesions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Egyptian patients with OLP
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-08-22 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
prolactin receptors expression in oral mucous membrane | 24 hours
  immuno-histochemistry

CONTACTS AND LOCATIONS:
Locations (1):
- October University for modern sciences and arts, Giza, Egypt